CLINICAL TRIAL: NCT06766240
Title: the Role of MRI in Evaluation of Low Back Pain in Middle Aged Females
Brief Title: the Role of MRI in Evaluation of Low Back Pain
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Safia Rafaat Mohamed, Resident, Diagnostic and Interventional Radiology department, Sohag University Hospital, Sohag University., Sohag University
Other Study IDs: Soh-Med-24-11-08MS
Record Dates: First submitted 2024-12-29; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- femles with low back pain: middle aged female patients aged from 40 to 60 years with complaint of low back pain who were referred to the department of radiology of sohag university hospital for Lumbosacral spine MRI. MRI imaging using Philips Achieva1.5T MRI device (Philips Achieva, Netherlands) or Siemens Magnetom Altea1.5T MRI device (Siemens Healthineers, Germany). the sequences used are Axial T2W; Sagittal T1W, T2W, Sagittal STIR, Coronal STIR and post gadolinium if needed.
  Interventions: Device: MRI on lumbosacral spine

INTERVENTIONS:
Device: MRI on lumbosacral spine — MRI imaging on lumbosacral spine using Philips Achieva1.5T MRI device (Philips Achieva, Netherlands) or Siemens Magnetom Altea1.5T MRI device (Siemens Healthineers, Germany). the sequences used are Axial T2W; Sagittal T1W, T2W, Sagittal STIR, Coronal STIR and post gadolinium if needed.

SUMMARY:
This study aims to evaluate the role of MRI to diagnose different causes of low back pain among middle aged females at Sohag university hospital.

ELIGIBILITY:
Inclusion Criteria:

- middle aged female patients aged from 40 to 60 years with complaints of low back pain who were referred to the department of radiology of sohag university hospital for Lumbosacral spine MRI.

Exclusion Criteria:

* Male patients.
* female patients aged less than 40 years or more than 60 years.
* Contraindication to magnetic resonance imaging including cochlear implant, pacemaker, claustrophobia.
* Non-cooperative sick patients.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: middle aged females complaining of low back pain in Sohag.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-06-12 (Estimated); Study Completion 2025-06-12 (Estimated)

PRIMARY OUTCOMES:
Magnetic Resonance Imaging (MRI) for diagnosis of low back pain in middle aged females | 6 months postmenopausal
  disc degeneration

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

REFERENCES:
- [Background] Bailey A. Risk factors for low back pain in women: still more questions to be answered. Menopause. 2009 Jan-Feb;16(1):3-4. doi: 10.1097/gme.0b013e31818e10a7. No abstract available. PMID 19002014
- [Background] Chou R, Fu R, Carrino JA, Deyo RA. Imaging strategies for low-back pain: systematic review and meta-analysis. Lancet. 2009 Feb 7;373(9662):463-72. doi: 10.1016/S0140-6736(09)60172-0. PMID 19200918
- [Background] Cousins JP, Haughton VM. Magnetic resonance imaging of the spine. J Am Acad Orthop Surg. 2009 Jan;17(1):22-30. doi: 10.5435/00124635-200901000-00004. PMID 19136424